CLINICAL TRIAL: NCT05627284
Title: A Prospective Clinical Trial of Colostomy-replacement Combined With Bio-mesh Placement in the Prevention of SSIH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-LCYJ-PY-33
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-10

CONDITIONS: Stoma Site Incisional Hernia
Keywords: Stoma Site Incisional Hernia; Colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stoma reversal with bio-mesh placement (Experimental)
  Interventions: Procedure: Stoma reversal with bio-mesh placement

INTERVENTIONS:
Procedure: Stoma reversal with bio-mesh placement — Patients will receive stoma reversal. During the surgery, a bio-mesh is placed beyond the peritoneum on the surgical site to strengthen the abdominal wall.

SUMMARY:
The goal of this clinical trial is to explore the safety and effectiveness of stoma reversal combining bio-mesh placement in patients with high risk of stoma site incisional hernia (SSIH). The main questions it aims to answer are:

* Whether bio-mesh placement is safe for patients with a high risk of SSIH.
* Whether stoma reversal combining bio-mesh placement is a preventive strategy for patients with high risk of SSIH.
* Whether stoma reversal combining bio-mesh placement will trigger other complications.

Participants who are eligible and are enrolled in this study will receive stoma reversal combining bio-mesh placement surgery. After that, they will be followed up for one year to evaluate the occurrence of SSIH and other complications.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old;
* Patients should have colonic prophylactic stoma and have not received reversal yet;
* There are no obvious signs of tumor recurrence or metastasis in tumor patients before stoma resection;
* No serious underlying diseases, can tolerate general anesthesia surgery
* Preoperative ECOG (Eastern Cooperative Oncology Group) physical status score 0/1;
* Preoperative ASA (American Society of Anesthesiologists) grade I-III;
* Without vital organs function failure;
* All patients and their families signed informed consent before surgery.

Exclusion Criteria:

* Incapacitated persons;
* With a history of other types of hernia;
* Those who have had hernia mesh implantation before;
* Those who are allergic to bio-mesh or their components before;
* Combined with other surgeries;
* Severe mental illness;
* Severe respiratory disease;
* Severe liver and kidney insufficiency;
* Those who have absolute contraindications to surgery;
* Suffering from severe bleeding disorders or obvious abnormal coagulation function;
* History of unstable angina or myocardial infarction within 6 months;
* History of cerebral infarction or cerebral hemorrhage within 6 months;
* Continuous intravenous application of glucocorticoid within 1 month;
* The patient has participated or is participating in other clinical studies (within 6 months).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
stoma site incisional hernia | one-year after surgery
  Hernia occurs on the primary stoma site

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China